CLINICAL TRIAL: NCT01192828
Title: Oxidative Stress Markers In Inherited Homocystinuria And The Impact Of Taurine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-1376; FDR003907 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Homocystinuria
Keywords: cystathionine beta-synthase (CBS)
MeSH Terms: conditions — Homocystinuria | interventions — Taurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Taurine (Experimental): Treatment with Taurine
  Interventions: Drug: taurine

INTERVENTIONS:
Drug: taurine — Take Taurine for 4 1/2 days, two doses per day
  Other Names: Not Applicable. No other names.

SUMMARY:
Cystathionine beta-synthase deficiency is an inherited disease that results in elevation of a substance called homocysteine (Hcy) in blood and urine. Individuals with this disorder have a very high risk for developing blood clots and are at risk for developing eye and bone abnormalities. Current treatments are generally difficult to follow and can fail. Development of additional therapies has been limited by lack of understanding of how the disease works.

The purpose of this study is to see if oxidative stress and inflammation are involved in the disease process and if short-term supplementation with taurine is an effective treatment.

Funding source: FDA.

DETAILED DESCRIPTION:
Cystathionine beta-synthase deficient homocystinuria(CBSDH) is an inherited disease that results in elevation of a substance called homocysteine(Hcy)in blood and urine. Individuals with this disorder have a very high risk for developing blood clots that can cause a stroke or other life-threatening problems. In addition, these individuals have bone and joint tissue abnormalities.

Current treatment with an extremely strict diet and medication (betaine) is very difficult to follow, and often fails. Development of additional treatment strategies has been limited by a lack of knowledge and understanding of how this disease works. Hence, there is a need to better understand what causes the blood clots and the bone and joint tissue abnormalities.

New data suggest that oxidative stress and inflammation play a central role in animals with this disease. Limited data on humans with this disease support this as well. Further, data from animals with this disease suggests that taurine, a natural body substance and food product, which is low in these patients, mitigates this effect. This study is designed to follow-up on these data.

The purpose of the study is to increase our understanding of the disease process in this disorder, and to see in a pilot study if short-term supplementation with taurine is an effective intervention. The aims of the study are to:

1. see if substances (markers) associated with oxidative stress and inflammation are increased in individuals with CBSDH
2. see if the levels of these markers relate to the levels of homocysteine
3. see if the levels of these markers decrease with short-term taurine supplementation
4. see how bood vessels and platelets (small substances in the blood that help blood clot) work in individuals with CBSDH, if their ability to work is related to levels of markers of oxidative stress and inflammation, and if taurine supplementation improves how they work
5. see if alterations of bone strength are related to levels of markers of inflammation.

The hypotheses to be investigated are as follows:

* Biomarkers of oxidative stress and inflammation are increased in individuals with CBSDH
* The degree of elevation of the biomarkers of oxidative stress and inflammation is relative to the degree of elevation of homocysteine, the main accumulating substance for this disease.
* Treatment with taurine mitigates the elevation of biomarkers of oxidative stress and inflammation.
* Endothelial function (blood vessel function) is abnormal in individuals with CBSDH even when receiving standard therapy and is improved with taurine supplementation.
* Chronic platelet aggregation, a variable finding in individuals with CBSDH, is mitigated with taurine supplementation.
* Decreased bone mineral density relates to the increase in inflammatory markers in CBSDH.

In addition, baseline pharmacokinetics (how much taurine is in the blood) of oral pharmacologic doses of taurine will be developed.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed biochemical, molecular, or enzymatic diagnosis of classic homocystinuria due to cystathionine beta-synthase deficiency (OMIM 236200)
2. And not fully responsive to therapy (eg, total homocysteine (tHcy) levels above 50 µmol/L on therapy including on B6 therapy)
3. Be over 8 years old and less than 50 years. The first four patients will be adults (age 18-50 years)
4. Be able and willing to provide informed consent

Exclusion Criteria:

1. Pregnancy: Females who are pregnant or lactating will be excluded from the study as the influence of pregnancy on the markers is not known nor is the safety of taurine supplementation in pregnancy.
2. Continued antioxidant intake:

   1. Individuals currently taking taurine, over the counter energy drinks containing taurine or other high dose antioxidants and unwilling to discontinue this for the study period (including a 2 week wash out period) will be excluded as such intake will likely impact laboratory results.
   2. Individuals taking Vitamin C as a prescribed treatment for their homocystinuria will be excluded as the antioxidant therapy may impact antioxidant and inflammation markers. (As Vitamin C is not standard of care for this disease we anticipate this to have minimal impact on recruitment.)
   3. Individuals currently taking platelet aggregation inhibitors such as salicylate on a self prescribed basis and unwilling to discontinue this for the study period (including a washout period of at least two weeks prior to the study) will be excluded as salicylate intake will impact platelet study results. Individuals taking salicylate (or other platelet aggregation inhibitors) prescribed as a therapy for their homocystinuria or other health issues will not be asked to stop the medication. They will participate in the study, but will be excluded only from the platelet studies.
3. Medication interactions: Individuals unable or unwilling to abstain from use of cyclic guanosine monophosphate (cGMP) phosphodiesterase 5 inhibitors (such as Viagra) during the study period will be excluded from the nitroglycerin-induced flow-mediated dilatation studies in accordance with known labeling contraindications.
4. Inflammatory status:

   1. Individuals who have a significant chronic illness that has a marked inflammatory component will be excluded from the study as the illness will impact inflammatory markers.
   2. Patients with an acute illness, which may impact inflammatory biomarkers, will be postponed for study entry until the acute illness is resolved. Entry into the study at a later day will be offered.
5. Recent cardiovascular event. Cardiovascular events (stroke, myocardial infarct, deep vein thrombosis, pulmonary embolus, thrombosis, or uncontrolled hypertension) may interfere with platelet function studies and with various mediators during the first months after the event. Patients who had such an event within the last 6 months will be excluded.
6. Hypertriglyceridemia. Individuals with a triglyceride level above 300 mg/dl will be excluded from the study.
7. Informed consent: Individuals who are unwilling or unable to consent, or in the case of minors who are unwilling or unable to assent will be excluded due to lack of ability to ensure informed consent.
8. Study compliance and integrity: Individual who anticipate an inability to comply with study procedures and requirements will be excluded.

   -

Ages: 8 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan VanHove, MD PhD MBA, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - Childrens Hospital Colorado, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - Duke University, Durham, North Carolina
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and recruited from three sites in the United States.
Pre-assignment Details: After enrollment a washout period for medications was required. At first study visit, assignment to arm occurred. One individual, while consented, did not participate at first study visit due to acute illness, was never rescheduled, and was removed. Number of subjects who started arm and completed study was thus 14.
Groups:
- Taurine Intervention: For safety reason, the first two subjects studies received low dose taurine therapy: 25 mg/kg body weight twice a day (maximum dose 1.5 grams). The next subjects received target high dose therapy: 75 mg/kg body weight twice a day (maximum dose of 5 grams).
Period: Overall Study
Arm/Group | Taurine Intervention
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Taurine Intervention: Treatment with taurine for 4 1/2 days, two doses per day
Arm/Group | Taurine Intervention
Number analyzed (Participants) | 14
Age, Customized [Count of Participants; unit: Participants] — Population: Total number of participant enrolled in study was 15. One subject who enrolled per phone had to postpone study visit due to acute illness. This individual failed to reschedule for study visit and was eventually removed from the study. Number of subjects who completed study and analyzed is therefore 14.
  Participants
    Age Distribution by Meaningful Groups: Prepubertal (8-12 years) | 4
    Age Distribution by Meaningful Groups: Teenagers (12-<20 years) | 4
    Age Distribution by Meaningful Groups: Young Adults (20-<30 years) | 4
    Age Distribution by Meaningful Groups: Older Adults (30-50 years) | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Total number of participant enrolled in study was 15. One subject who enrolled per phone had to postpone study visit due to acute illness. This individual failed to reschedule for study visit and was eventually removed from the study. Number of subjects who completed study and analyzed is therefore 14.
  Participants
    Female | 6
    Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Total number of participant enrolled in study was 15. One subject who enrolled per phone had to postpone study visit due to acute illness. This individual failed to reschedule for study visit and was eventually removed from the study. Number of subjects who completed study and analyzed is therefore 14
  Participants
    Categories: Native American | 0
    Categories: Asian | 0
    Categories: Black | 2
    Categories: White | 9
    Categories: Hispanic | 3
    Categories: Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference in Thiobarbituric Acid Reactive Substances (TBARS) in Individuals With Cystathionine Beta Synthase Deficient Homocystinuria (CBSDH) Pre and Post Taurine Treatment.
Description: TBARS were measured in plasma via colorimetric absorbance. TBARS are a marker of oxidative stress. They are formed as a by-product of lipid (fat) oxidation. TBARS predominantly reflect the level of malondialdehyde (MDA) a substance that is formed from the breakdown of polyunsaturated fatty acids.
Time Frame: Baseline and after 4 days of therapy.
Population: Analyzable data from all individuals with CBSDH who received the target dose of taurine were used for the calculations. The two individuals treated with low dose taurine were excluded from he analysis.
Measure: Mean (Standard Error); unit: nmol/ml
Groups:
- Taurine Intervention Group: For safety reason, the first two subjects studies received low dose taurine therapy: 25 mg/kg body weight twice a day (maximum dose 1.5 grams). There after all received target dose therapy: 75 mg/kg body weight twice a day (maximum dose of 5 grams).
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 12
nmol/ml
  Pre Treatment | 3.47 (0.18)
  Post treatment | 3.16 (0.27)
Statistical Analysis 1: Comparison: Taurine Intervention Group; Null hypothesis applied; Test type: Other — Descriptive analysis; p = 0.235, t-test, 2 sided; paired

2. Primary Outcome: Difference in Tumor Necrosis Factor Alpha (TNF-alpha) in Individuals With CBSDH Pre and Post Taurine Treatment.
Description: TNF-alpha was measured in plasma via Luminex high sensitivity assay. TNF-alpha is a signaling protein, or cytokine that promotes an inflammatory response.
Time Frame: Baseline and after 4 days of treatment.
Population: Analyzable data from all individuals with CBSDH who received the target dose of taurine were used for the calculations. The two individuals treated with low dose taurine were excluded from the analysis.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 12
pg/ml
  Pre treatment | 5.95 (0.39)
  Post treatment | 6.07 (0.49)
Statistical Analysis 1: Comparison: Taurine Intervention Group; Null hypothesis assumed; Test type: Other — Descriptive analysis; p = 0.701, t-test, 2 sided; paired

3. Secondary Outcome: Difference in Endothelial Function (Blood Vessel Function) in Individuals With CBSDH Pre and Post Taurine Treatment
Description: Endothelial function was measured by doppler brachial artery flow-mediated dilation (FMD) studies.
Time Frame: Baseline and after 4.5 days of taurine treatment
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mm
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 12
mm
  Pre treatment | 9.80 (1.76)
  Post treatment | 11.57 (1.21)
Statistical Analysis 1: Comparison: Taurine Intervention Group; Null hypothesis applied; Test type: Other — Descriptive analysis; p = 0.190, t-test, 2 sided; paired t-test

4. Secondary Outcome: Difference in Endothelial Function (Blood Vessel Function) in Individuals With CBSDH and Homocysteine Levels Greater Than 125 Micromole/L Pre and Post Taurine Treatment.
Description: Endothelial function was measured by doppler brachial artery flow-mediated dilation (FMD) studies.
Time Frame: Baseline and after 4.5 days of therapy.
Population: Analyzable data from all individuals with CBSDH having baseline homocysteine levels greater than 125 micromole/L who received the target dose of taurine were used for the calculations. The two individuals treated with low dose taurine were excluded from the analysis.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 6
mm
  Pre treatment | 7.25 (1.23)
  Post treatment | 11.10 (1.48)
Statistical Analysis 1: Comparison: Taurine Intervention Group; Null hypothesis applied; Test type: Other — Descriptive analysis; p = 0.052, t-test, 2 sided; paired t-test

5. Secondary Outcome: Difference in Endothelial Function (Blood Vessel Function) in Individuals With CBSDH and Pre Taurine Exposure FMD Values Less Than 10 mm Pre and Post Taurine Treatment.
Description: Endothelial function was measured by doppler brachial artery flow-mediated dilation (FMD) studies.
Time Frame: Baseline and after 4.5 days of therapy.
Population: Analyzable data from all individuals with CBSDH studied with baseline flow mediated dilation values of less than 10 mm and who received the target dose of taurine were used for the calculations. The two individuals treated with low dose taurine were excluded from the analysis.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 8
mm
  Pre Treatment | 5.98 (0.51)
  Post Treatment | 9.86 (1.28)
Statistical Analysis 1: Comparison: Taurine Intervention Group; Null hypothesis assumed; Test type: Other — Descriptive analysis; p = 0.014, t-test, 2 sided; paired t-test

6. Secondary Outcome: Percent of Individuals With Decreased Bone Mineral Density.
Description: Bone mineral density was assessed via whole body dual energy X-ray absorptiometry (DEXA) with bone density corrected for age. The absolute DEXA value was not used for analysis, rather values below 2 standard deviations of normal were taken as evidence of osteoporosis.
Time Frame: Baseline
Population: Analysis was on all analyzable data from subjects with CBSDH who participated in the active study and data from control population as provided by DEXA report.
Measure: Count of Participants; unit: Participants
Groups:
- Taurine Intervention: Baseline value prior to taurine intervention.
Arm/Group | Taurine Intervention
Number analyzed (Participants) | 14
Participants
  Normal bone mineral denisty | 14
  Abnormal bone mineral density | 0

7. Other Pre Specified Outcome: Thiobarbituric Acid Reactive Substances (TBARS) in Individuals With CBSDH Compare to Homocysteine Level.
Description: TBARS were measured in plasma via colorimetric absorbance. Homocysteine was measured in serum by gas chromatography/mass spectrometry (GC/MS) in a Clinical Laboratory Improvements Amendments (CLIA) approved clinical laboratory. TBARS are a marker of oxidative stress. TBARS are formed as a by-product of lipid (fat) oxidation. TBARS predominantly reflect the level of malondialdehyde (MDA) a substance that is formed from the breakdown of polyunsaturated fatty acids.
Time Frame: Baseline
Population: Analyzable data from all subjects with CBSDH who completed day one of active study and normal homocysteine values provided by assaying laboratory were used for the calculations.
Measure: Mean (Standard Error); unit: micromol/l
Groups:
- Taurine Intervention Group: Baseline value prior to taurine intervention on day two of study.
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 14
micromol/l
  TBARS | 0.00365 (0.00087)
  Homocysteine | 161 (67.2)
Statistical Analysis 1: Comparison: Taurine Intervention Group; Null hypothesis assumed; Test type: Other — Descriptive analysis; p = .541, Spearman's rank correlation; Spearman's rank correlation rho is 0.179, with p value 0.541, N is 14

8. Other Pre Specified Outcome: Determination of Baseline Taurine Level, Peak Taurine Level on Day One, Trough Level on Day One and Trough Level on Day Four of Taurine Treatment.
Description: Taurine was measured in plasma via liquid chromatogram(LC)-MS/MS.
Time Frame: Taurine levels were obtained prior to taurine adminstration and at , t=0.5, t=1, t=2, t=3, t=4, t=6, t=8, t=12 and 96 hours.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microM
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 12
microM
  Baseline value | 40.5 (11.9)
  Peak Value Day One | 753.0 (240.0)
  Trough Value Day One 12h | 50.0 (14.0)
  Trough Value Day Four | 82.0 (36.2)

9. Other Pre Specified Outcome: Difference in Triglycerides in Individuals With CBSDH Receiving Both Low Dose and Target Dose Taurine Pre and Post Taurine Treatment (Safety Assessment)
Description: Triglycerides were measured in a CLIA approved clinical laboratory.Triglycerides are a natural occurring fat. High levels over a long period of time can increase the chances for heart disease. Levels greater that 1000 mg/dl over a short period of time can increase chances of pancreatitis.
Time Frame: Baseline and after 4 days of treatment.
Population: Analyzable data from all individuals with CBSDH who were treated with taurine, this being both low dose and targeted dose of medication.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 14
mg/dL
  Pre Taurine | 77.5 (19.0)
  Post Taurine | 116.7 (33.4)
Statistical Analysis 1: Comparison: Taurine Intervention Group; Null hypothesis assumed; Test type: Other — Descriptive analysis; p = 0.014, t-test, 2 sided; paired t-test

10. Other Pre Specified Outcome: Difference in Triglycerides in Individuals With CBSDH Receiving Target Dose Taurine Pre and Post Taurine Treatment (Safety Assessment)
Description: Triglycerides were measured in a CLIA approved clinical laboratory. Triglycerides are a natural occurring fat, High levels over a long period of time can increase the chances for heart disease. Levels greater that 1000 mg/dl over a short period of time can increase chances of pancreatitis.
Time Frame: Baseline and after 4 days of treatment.
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 12
mg/dL
  Pre Treatment | 61.6 (12.7)
  Post Treatment | 98.7 (29.7)
Statistical Analysis 1: Comparison: Taurine Intervention Group; Null hypothesis assumed; Test type: Other — Descriptive analysis; p = 0.012, t-test, 2 sided; paired t-test

11. Other Pre Specified Outcome: Difference in Systolic Blood Pressure in Individuals With CBSDH Receiving Both Low Dose and Target Dose Taurine Pre and Post Taurine Treatment (Safety Assessment).
Time Frame: Baseline and after 4 days of treatment.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 14
mmHg
  Pre Taurine | 116 (12)
  Post Taurine | 112 (12)
Statistical Analysis 1: Comparison: Taurine Intervention Group; Null hypothesis applied; Test type: Other — Descriptive analysis; p = 0.160, t-test, 2 sided; paired t-test

12. Other Pre Specified Outcome: Difference in Diastolic Blood Pressure in Individuals With CBSDH Receiving Both Low Dose and Target Dose Taurine Pre and Post Taurine Treatment (Safety Assessment).
Time Frame: Baseline and after 4 days of treatment.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Taurine Intervention Group
Number analyzed (Participants) | 14
mmHg
  Pre Taurine | 70 (10)
  Post Taurine | 68 (8)
Statistical Analysis 1: Comparison: Taurine Intervention Group; Test type: Other — Descriptive analysis; p = 0.10, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 19 days (During the 5 days taurine was administered plus two weeks after taurine administration.)
Groups:
- Taurine Intervention: Taurine Intervention
Arm/Group | Taurine Intervention
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 5/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taurine Intervention (N=14)
Gastrointestinal symptoms (Gastrointestinal disorders) | 5 (6)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT01192828/Prot_SAP_000.pdf